CLINICAL TRIAL: NCT02970032
Title: Evaluation of Anti-Xa Levels in Surgery Patients Receiving Fixed Dose Heparin
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Corinne Bertolaccini, Pharmacist, University of Utah
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB_00095514
Record Dates: First submitted 2016-11-11; First posted 2016-11-21 (Estimated); Results first posted 2019-06-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Deep-Venous Thrombosis; Pulmonary Embolism; Venous Thromboembolism
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard heparin dose (Active Comparator): The investigators will identify surgical patients placed on fixed dose heparin infusions at their attending surgeon's discretion-the proposed research will not dictate the initiation of the heparin drip intraoperatively. However, the investigators will identify patients already on heparin, evaluate steady state heparin anti-Xa levels and adjust patient's dose if necessary based on steady state anti-Xa levels. Eligible patients will be started on heparin fixed-dose intraoperatively. Steady state anti-Xa levels will be drawn at least 6 hours after initiation of heparin infusion. Goal anti-Xa levels will be 0.1-0.35 IU/mL.
  Interventions: Drug: Standard heparin dose
- Real time heparin dose adjustment (Experimental): Patients with identified out of range levels will receive pharmacist-driven real time heparin dose adjustment and will receive follow-up steady state anti-Xa levels. Anti-Xa level monitoring will be discontinued when in range peak levels are obtained, when heparin infusions are discontinued at surgeon discretion, or when the patient is discharged.
  Interventions: Drug: Real time heparin dose adjustment

INTERVENTIONS:
Drug: Real time heparin dose adjustment — Patients will have steady state anti-Xa levels drawn at least 6 hours after initiation of heparin infusion. Patients with out of range anti-Xa levels will receive real time heparin dose adjustment followed by repeat anti-Xa levels.
  Arms: Real time heparin dose adjustment
Drug: Standard heparin dose — Patients will be placed on heparin infusions per their surgeon's discretion.
  Arms: Standard heparin dose

SUMMARY:
The purpose of this study is to determine if fixed dose heparin infusions at a rate of 500 units/hour are sufficient to maintain a target anti-Xa of 0.1-0.35 IU/mL for venous thromboembolism (VTE) prophylaxis in patients undergoing microvascular surgery. Additionally, a pilot protocol has been developed to titrate these heparin infusions to ensure patients have sufficient VTE prophylaxis. All patients will be enrolled in the observational arm of the study and receive anti-Xa level monitoring. Patients with out-of-range anti-Xa levels will cross over to the interventional arm of the study and receive real time heparin infusion dose adjustments per the pilot protocol. The primary outcome measured will be the percentage of patients with anti-Xa levels in the target range of 0.1-0.35 IU/mL while on a heparin infusion at 500 units/hour.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgical procedures
* Initiation of a heparin infusion at a rate of 500 units/hour intraoperatively or postoperatively

Exclusion Criteria:

* Age <18 years old
* Pregnant
* Incarcerated
* Mentally disabled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2017-09-10 (Actual); Study Completion 2017-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Bertolaccini, PharmD, Principal Investigator — University of Utah Health
Locations (1):
- Univeristy of Utah Hospital, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All 20 patients that were enrolled in the standard heparin dose arm crossed over into the real time heparin dose adjustment arm per the pilot protocol with undetectable anti-Xa levels (<0.10).
Groups:
- Standard Heparin Dose Followed by Dose Adjustment: The investigators will identify surgical patients placed on fixed dose heparin infusions at their attending surgeon's discretion-the proposed research will not dictate the initiation of the heparin drip intraoperatively. However, the investigators will identify patients already on heparin, evaluate steady state heparin anti-Xa levels and adjust patient's dose if necessary based on steady state anti-Xa levels. Eligible patients will be started on heparin fixed-dose intraoperatively. Steady state anti-Xa levels will be drawn at least 6 hours after initiation of heparin infusion. Goal anti-Xa levels will be 0.1-0.35 IU/mL.
  Patients with identified out of range levels will receive pharmacist-driven real time heparin dose adjustment and will receive follow-up steady state anti-Xa levels. Anti-Xa level monitoring will be discontinued when in range peak levels are obtained, when heparin infusions are discontinued at surgeon discretion, or when the patient is discharged.
Period: Standard Heparin Dose
Arm/Group | Standard Heparin Dose Followed by Dose Adjustment
Started | 20
Completed | 20
Not Completed | 0
Period: Real Time Heparin Dose Adjustment
Arm/Group | Standard Heparin Dose Followed by Dose Adjustment
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Heparin Dose Followed by Dose Adjustment: The investigators will identify surgical patients placed on fixed dose heparin infusions at their attending surgeon's discretion-the proposed research will not dictate the initiation of the heparin drip intraoperatively. However, the investigators will identify patients already on heparin, evaluate steady state heparin anti-Xa levels and adjust patient's dose if necessary based on steady state anti-Xa levels.Steady state anti-Xa levels will be drawn at least 6 hours after initiation of heparin infusion. Goal anti-Xa levels will be 0.1-0.35 IU/mL. Patients with identified out of range levels will receive pharmacist-driven real time heparin dose adjustment and will receive follow-up steady state anti-Xa levels. Anti-Xa level monitoring will be discontinued when in range peak levels are obtained, when heparin infusions are discontinued at surgeon discretion, or when the patient is discharged.
Arm/Group | Standard Heparin Dose Followed by Dose Adjustment
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Number; unit: Kilograms] | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Anti-Xa Levels Within Target Range (0.1-0.35 IU/mL)
Description: Anti-Xa levels are used to monitor anticoagulant therapy.
Time Frame: Through study completion, an average of 1 year.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Heparin Dose Followed by Dose Adjustment
Number analyzed (Participants) | 20
Participants
  Standard Heparin Dose | 0
  Dose adjustment | 12

2. Secondary Outcome: Number of Rate Adjustments
Description: Heparin rate adjustments were made for out of range anti-Xa levels (<0.1 and >0.35)
Time Frame: Through study completion, an average of 1 year.
Population: During the dose adjustment period, anti-Xa levels were monitored and dose adjustments made per the pilot protocol.
Measure: Mean (Full Range); unit: Rate adjustments
Arm/Group | Standard Heparin Dose Followed by Dose Adjustment
Number analyzed (Participants) | 20
Rate adjustments | 4.5 [1 to 9]

ADVERSE EVENTS:
Time Frame: 3 months from discharge
Arm/Group | Standard Heparin Dose | Real Time Heparin Dose Adjustment
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/20
Other Adverse Events (participants affected / at risk) | 1/20 | 1/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Heparin Dose (N=20) | Real Time Heparin Dose Adjustment (N=20)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Heparin Dose (N=20) | Real Time Heparin Dose Adjustment (N=20)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-24): https://cdn.clinicaltrials.gov/large-docs/32/NCT02970032/Prot_SAP_000.pdf